CLINICAL TRIAL: NCT00266292
Title: The Effect of n-3 LCPUFA on Immune Function and Cardiovascular Risk Factors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Copenhagen (Other)
Collaborators: Danish Research Agency (Other); Hjerteforeningen (Unknown); Technical University of Denmark (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: KF 01 267804; SJVF 23-04-0050; IHE project no. A-304
Record Dates: First submitted 2005-12-15; First posted 2005-12-16 (Estimated); Last update posted 2010-05-28 (Estimated); Status verified 2005-12

CONDITIONS: Cardiovascular Heart Disease; Metabolic Syndrome
Keywords: Fish oil; Polyunsaturated fatty acid; Immune function; Endothelial function; Cardiovascular risk factors
MeSH Terms: conditions — Metabolic Syndrome | interventions — Fish Oils

INTERVENTIONS:
Behavioral: Fish oil (Bio-Marine, Pharma Nord)
Behavioral: n-6 PUFA intake (Margarine+sunflower oil vs. butter product+rapeseed oil)

SUMMARY:
The purpose of this study is to investigate the effects of long-chain n-3 polyunsaturated fatty acids (n-3 LCPUFA) on immune function and cardiovascular disease risk

DETAILED DESCRIPTION:
In a controlled, double-blinded human intervention study the effects of fish oil versus control (olive oil) and of a high versus low consumption of n-6 polyunsaturated fatty acids are investigated. Sixty-seventy healthy men will be randomized to oil capsules and to substitute their dietary fats with one of two types of oil and butter-product that we provide. Outcome variables are ex vivo cytokine production in full blood and isolated immune cells after 24 h of stimulation with bacteria or bacterial components, blood pressure and arterial function, plasma concentrations of cholesterol, triacylglycerol, C-reactive protein and a number of other markers of endothelial function and cardiovascular risk.

The hypotheses are that both increased intake of n-3 polyunsaturated fatty acids (from fish oil) and a low consumption of n-6 polyunsaturated fatty acids increase incorporation of docosahexanoic acid in immune cell membranes and that this decreases the inflammatory response and potential and improve overall cardiovascular disease risk.

The mechanistic aspects of this will be further explored by in vitro studies with monocytes cultured in the presence of varying amounts of polyunsaturated fatty acids.

ELIGIBILITY:
Inclusion Criteria:

* Healthy (no chronic diseases and no regular medications)
* BMI >18.5 and <27.5 kg/m2
* Daily use of fats and home cooking >5 d/wk
* Heavy exercise <7 h/wk
* Not daily smokers (<5 cigarets/wk)

Exclusion Criteria:

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60
Dates: Start 2005-09; Study Completion 2006-04

PRIMARY OUTCOMES:
Fatty acid composition of PMBC - before and after 2 mo of interventions and after 2 mo of follow-up
Ex vivo cytokine production (e.g. IL-6, TNF-α, IL-10, and interferon-γ) in whole blood and PBMC cultures after 24 h of stimulation - before and after interventions and after follow up
Plasma CRP, IL-6 & fibrinogen - before, after and follow-up
Plasma lipid profile: TAG, cholesterol, LDL & HDL - before, after and follow-up
Blood pressure - before, after and follow-up

SECONDARY OUTCOMES:
Anthropometric measures - before, after & follow-up
Ex vivo cytokine production in isolated monocytes - after intervention only
Endothelial function (PWV and/or arterial compliance) - before & after
Superoxide production in full blood samples - before & after
Plasma insulin/glucose - before, after and follow-up
Plasma markers of endothelial function (e.g. VCAM-1, ICAM-1, Matrix metallo proteinases, E- & P-selectin, nitrite and endothelin-1) - before and after
Plasma CD40L - before, after and follow-up
RBC fatty acid composition - before, after and follow-up
Coagulation factors (e.g. PAI, tPA, factor VII) - before, after and follow-up
Folate/homocysteine - before. after and follow-up
Lipoprotein(a) - before, after and follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Lotte Lauritzen, Ph.D, Principal Investigator — Department of Human Nutrition, Royal Veterinary and Agricultural University, Denmark
Locations (1):
- Department of Human Nutrition, Frederiksberg, Denmark

REFERENCES:
- [Result] Damsgaard CT, Lauritzen L, Calder PC, Kjaer TR, Frokiaer H. Reduced ex vivo interleukin-6 production by dietary fish oil is not modified by linoleic acid intake in healthy men. J Nutr. 2009 Jul;139(7):1410-4. doi: 10.3945/jn.108.102269. Epub 2009 Jun 3. PMID 19494025
- [Result] Damsgaard CT, Lauritzen L, Calder PC, Kjaer TM, Frokiaer H. Whole-blood culture is a valid low-cost method to measure monocytic cytokines - a comparison of cytokine production in cultures of human whole-blood, mononuclear cells and monocytes. J Immunol Methods. 2009 Jan 30;340(2):95-101. doi: 10.1016/j.jim.2008.10.005. Epub 2008 Nov 8. PMID 19000693
- [Result] Damsgaard CT, Frokiaer H, Andersen AD, Lauritzen L. Fish oil in combination with high or low intakes of linoleic acid lowers plasma triacylglycerols but does not affect other cardiovascular risk markers in healthy men. J Nutr. 2008 Jun;138(6):1061-6. doi: 10.1093/jn/138.6.1061. PMID 18492834
- [Result] Bartelt S, Timm M, Damsgaard CT, Hansen EW, Hansen HS, Lauritzen L. The effect of dietary fish oil-supplementation to healthy young men on oxidative burst measured by whole blood chemiluminescence. Br J Nutr. 2008 Jun;99(6):1230-8. doi: 10.1017/S0007114507853451. Epub 2008 Jan 17. PMID 18199388